CLINICAL TRIAL: NCT02567292
Title: Effects of an Exclusive Human Milk Diet on Enteral Feeding Outcomes of Neonates With Congenital Gastrointestinal Disorders
Brief Title: Human Milk for Congenital Gastrointestinal Disorders
Acronym: HM for CGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Chatham Valley Foundation (Unknown); Prolacta Bioscience (Industry)
Responsible Party: Principal Investigator, Heidi Karpen, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00080481
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Congenital Gastrointestinal Disorders
Keywords: Digestive Disease and Disorders; Neonatal; Pediatric Disorders
MeSH Terms: conditions — Digestive System Diseases; Disease | interventions — Milk, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrospective Control Group (No Intervention): Approximately 150 patients with congenital gastrointestinal disorders who were treated in the neonatal intensive care unit (NICU) at Children's Healthcare of Atlanta-Egleston and other participating institutions from 2012 to 2015, who had non-human milk (HM) diets will be identified as retrospective controls using the electronic medical records system.
- Exclusive Human Milk Diet Group (Experimental): A minimum of 150 patients with CGD admitted to participating NICUs who meet inclusion criteria and provide informed consent will be enrolled in the prospective arm of the study. These patients will be fed an EHMD comprised of mother's own milk (MOM) or pasteurized donor human milk (DM). Fortification will be provided with human milk derived human milk fortifier, either a human milk-based fortifier (Prolact+ H2MF®) for infants born at less than 37 weeks GA or <2,200g birth weight or the term-equivalent version (PBCLN-002) formulated for infants >37 weeks and/or >2,200g at birth. Infants will receive this EHMD until they have achieved full enteral feedings for 7 days with bowel in continuity
  Interventions: Other: Human Milk

INTERVENTIONS:
Other: Human Milk — Participants will receive an exclusive human milk diet comprised of mother's own milk (MOM, pasteurized donor human milk (DM) fortified with a donor-milk based fortifier (DMBF): Prolact+ for infants <37 weeks PMA and/or or weight <2,200g or PBCLN-002 for infants >37 weeks PMA and/or weight >2,200g)
  Arms: Exclusive Human Milk Diet Group

SUMMARY:
This study aims to identify whether an exclusive human milk diet (EHMD) would improve outcomes in neonates with congenital gastrointestinal disorders (CGD) and by facilitating an earlier transition off of parenteral nutrition (PN).

DETAILED DESCRIPTION:
Infants born with congenital gastrointestinal disorders (CGD) can be very challenging to treat. The CGD require surgery shortly after birth to correct the problems and recovery can take a long time.

During the period of time the infant's intestines are sick or don't work properly, they rely on parenteral nutrition (IV fluids containing carbohydrates, proteins and fats) to meet their nutritional needs. Being on PN for a long time requires special intravenous lines, and increases the risk of blood stream infections and can make the liver sick.

Feeding babies who have these CGD is often very difficult, as the intestine needs to adapt. It needs to make appropriately formed stool to eliminate wastes, but not lose too much water or too many electrolytes. There is often a lot of starting and stopping of feeds. Human milk (HM) is considered the ideal source of nutrition for all infants.

This study aims to identify whether an exclusive human milk diet (EHMD) would improve outcomes in neonates with congenital gastrointestinal disorders (CGD) and by facilitating an earlier transition off of parenteral nutrition (PN).

ELIGIBILITY:
Inclusion Criteria:

1. Admission to participating NICU at less than 7 days of age
2. Birthweight >1250g and/or gestational age at birth >32 weeks
3. Less than 7 days of enteral feedings
4. Diagnosis of eligible primary "Congenital Gastointestinal Disorders" defined as: gastroschisis, omphalocele and intestinal atresias
5. Consent to the use of donor human milk products
6. Consent to participate in this study

Exclusion Criteria:

1. Admission to participating NICU at >7 days of age
2. Birthweight <1250g and/or gestational age <32 weeks
3. Diagnosis of non-eligible gastrointestinal disorders: congenital diaphragmatic hernia, midgut volvulus, Hirschsprung's disease, esophageal atresia, imperforate anus
4. Evidence of significant liver dysfunction at time of enrollment (direct bilirubin >4 and transaminases elevated more than 2 SD above upper limit of normal for age)
5. Liver malformations such as biliary atresia and choledochal cyst
6. Refusal of consent

Ages: 1 Minute to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Time to full enteral feeding | From birth to day of life full enteral feedings for 7 days is achieved (up to 30 days)
  The number of days to achieve full enteral feeding after the initial human milk feeding

SECONDARY OUTCOMES:
Number of days of parenteral nutrition | Through study completion, up to 1 year
  The total number of days parenteral nutrition is required.
Growth | Through study completion, up to 1 year
  Compare growth parameters (weight, length and head circumference) as daily g/kg/d and z-scores birth to discharge
Difference in conjugated bilirubin levels | From birth to day of life full enteral feedings for 7 days is achieved (up to 30 days)
  The difference in average bilirubin level will be compared between the non-human milk diet (retrospective control group) and the breast milk diet group.
Length of hospital stay | Through study completion, up to 6 months
  The length of hospital stay described as the number of days spent in the hospital
Feeding interruptions | From birth to day of life full enteral feedings for 7 days is achieved (up to 30 days)
  NPO for at least 24 hours. NPO due to elective surgeries or procedures will not be defined as feeding interruptions
Feeding intolerance | From birth to day of life full enteral feedings for 7 days is achieved (up to 30 days)
  Number of days when one or more feedings were held for clinical concerns
Episodes of Necrotizing Enterocolitis | From birth to day of life full enteral feedings for 7 days is achieved (up to 30 days)
  Number of episodes of Stage IIb NEC or greater
Number of sepsis episodes | From birth to day of life full enteral feedings for 7 days is achieved (up to 30 days)
  The number of sepsis episodes will be compared between the non-breast milk diet (retrospective control group) and the breast milk diet group.
Death rate | Through study completion, up to 1 year
  The number of deaths between participants who receive breast milk only diets as compared to the non-breast milk diet (retrospective control group while in the neonatal intensive care unit (NICU).

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Karpen, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta-Egleston, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shinnick JK, Wang E, Hulbert C, McCracken C, Sarson GY, Piazza A, Karpen H, Durham MM. Effects of a Breast Milk Diet on Enteral Feeding Outcomes of Neonates with Gastrointestinal Disorders. Breastfeed Med. 2016 Aug;11(6):286-292. doi: 10.1089/bfm.2016.0002. Epub 2016 Jun 22. PMID 27331420